CLINICAL TRIAL: NCT06173999
Title: A Phase Ib/II, Open-label, Multi-center Study of SHR2554 With CHOP/CHOEP in Treatment-naïve Patients With Peripheral T-cell Lymphoma
Brief Title: A Study of SHR2554 With Chemotherapy in Treatment-naïve Patients With Peripheral T-cell Lymphoma
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Jiangsu HengRui Medicine Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SHR2554-201
Record Dates: First submitted 2023-12-08; First posted 2023-12-18 (Actual); Last update posted 2024-05-14 (Actual); Status verified 2024-05

CONDITIONS: Peripheral T-cell Lymphoma
MeSH Terms: conditions — Lymphoma, T-Cell, Peripheral

STUDY DESIGN:
Intervention Model Description: SHR2554 with CHOP/CHOEP.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment group A (Experimental)
  Interventions: Drug: SHR2554/CHOP
- Treatment group B (Experimental)
  Interventions: Drug: SHR2554/CHOEP

INTERVENTIONS:
Drug: SHR2554/CHOP — SHR2554 with CHOP
  Arms: Treatment group A
Drug: SHR2554/CHOEP — SHR2554 with CHOEP
  Arms: Treatment group B

SUMMARY:
The study is being conducted to evaluate the safety and efficacy of SHR2554 with CHOP/CHOEP in treatment- naïve peripheral T-cell lymphoma.

ELIGIBILITY:
Inclusion Criteria:

1. Males or females aged 18-70 years (inclusive);
2. Histologically confirmed peripheral T-cell lymphoma;
3. Eastern Cooperative Oncology Group performance status (ECOG PS) score of 0 or 1;
4. Life expectancy ≥ 12 weeks;
5. Have measurable lesions ;
6. The subject is willing and able to comply with the visit schedule, dosing schedule, laboratory tests, and other clinical study procedures.

Exclusion Criteria:

1. Underwent major surgery or experienced severe trauma within 4 weeks prior to the first dose of the investigational drug;
2. Known active HBV or HCV infection;
3. History of clinically significant cardiovascular disease;
4. History of other malignancies within 5 years;
5. Pregnant or lactating women;
6. Based on the investigator's judgment, there are objective conditions that may prevent the subject from completing the study as planned or the subject has other factors, concomitant diseases, concomitant treatments, or abnormal laboratory findings that may lead to early study termination.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2023-12-22 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Safety endpoints: incidence and severity of adverse events (AEs) | through study completion, an average of about 6 months
  Ib phase
Overall response rate (ORR) | 90 days since the date of first dose
  II phase

SECONDARY OUTCOMES:
Plasma concentration | Day 1 of cycle 1 to day 1 of cycle 4 (21 days/cycle)
  Ib phase
Progression Free Survival (PFS) | through study completion, an average of about 6 months
  II phase
Overall Survival (OS) | 2 years since the date of first dose
  II phase
Duration of response (DOR) | through study completion, an average of about 6 months
  II phase
Incidence and severity of adverse events (AEs) | through study completion, an average of about 6 months
  II phase

CONTACTS AND LOCATIONS:
Locations (1):
- Beijing Cancer Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided